CLINICAL TRIAL: NCT00655785
Title: Phase Ｉ/Ⅱ Sturdy on Antiangiogenic Vaccine Therapy Using Epitope Peptide Derived From VEGFR1 and VEGFR2 With Gemcitabine in Treating Patients With Unresectable, Recurrent, or Metastatic Pancreatic Cancer
Brief Title: Antiangiogenic Peptide Vaccine Therapy With Gemcitabine in Treating Patient With Pancreatic Cancer (Phase1/2)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Fukushima Medical University (Other)
Collaborators: Human Genome Center, Institute of Medical Science, University of Tokyo (Other)
Responsible Party: Principal Investigator, Takashi Kimura, Assistant professor, Fukushima Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FPCR1R2-2
Record Dates: First submitted 2008-04-04; First posted 2008-04-10 (Estimated); Last update posted 2013-03-14 (Estimated); Status verified 2013-03

CONDITIONS: Pancreatic Cancer
Keywords: Epitope peptide; CTL; Pancreatic cancer; Vaccination VEGFR1; VEGFR2
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Phase 1/2 study (Experimental)
  Interventions: Biological: VEGFR1-1084, VEGFR2-169; Drug: Gemcitabine

INTERVENTIONS:
Biological: VEGFR1-1084, VEGFR2-169 — One mg of each peptide will be administered by subcutaneous injection on days 1, 8, 15, and 22 in group A, on days 3, 10, 17, 24 in group B, or 5, 12, 19, 26 in group C
Drug: Gemcitabine — Gemcitabine will be administered intravenously at a fixed dose of 1000mg/m2 on day 3, 10 and 17

SUMMARY:
The purpose of this study is to evaluate the safety, and tolerability of HLA-A*2402 restricted epitope peptide VEGFR1 and VEGFR2 emulsified with Montanide ISA 51 in combination with gemcitabine

DETAILED DESCRIPTION:
Vascular endothelial growth factor receptor 1 and 2 (VEGFR1 andVEGFR2) are essential targets to tumor angiogenesis, and we identified that peptides derived from these receptors significantly induce the effective tumor specific CTL response in vitro and in vivo. According to these findings, in this trial, we evaluate the safety, tolerability and immune response of these peptide emulsified with Montanide ISA 51 in combination with gemcitabine

ELIGIBILITY:
Inclusion Criteria:

DISEASE CHARACTERISTICS

1. Locally advanced or metastatic pancreatic cancer precluding curative surgical resection and recurrent pancreatic cancer
2. Measurable disease by CT scan

PATIENTS CHARACTERISTICS

1. ECOG performance status 0-2
2. Life expectancy > 3 months
3. Laboratory values as follows:

   * 2,000/mm3 < WBC < 15000/mm3
   * Platelet count ≥ 750,000/mm³
   * Total Bilirubin ≤ 1.5 x
   * Aspartate transaminase < 150 IU/L
   * Alanine transaminase < 150 IU/L
   * Creatinine ≤ 3.0 mg/dl
4. HLA-A*2402
5. Able and willing to give valid written informed consent

Exclusion Criteria:

1. Pregnancy (women of childbearing potential: Refusal or inability to use effective means of contraception)
2. Breast-feeder
3. Active or uncontrolled infection
4. Prior chemotherapy, radiation therapy, or immunotherapy within 4 weeks
5. Serious or uncured wound
6. Active or uncontrolled other malignancy
7. Steroids or immunosuppressing agent dependent status
8. Interstitial pneumonia
9. Ileus
10. Decision of unsuitableness by principal investigator or physician-in-charge

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2007-09; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
toxicities as assessed by NCI-CACAE ver3) | 3 months

SECONDARY OUTCOMES:
Differences of peptide specific CTL response in vitro among sequence of gemcitabine and peptide vaccine administration | 3months
CD8 population | 3months
Change in level of regulatory T cells | 3months
Objective response rate | 1year
feasibility | 1year
Survival | 1year

CONTACTS AND LOCATIONS:
Overall Officials: Mitsukazu Gotoh, M.D. & Ph.D, Study Chair — Fukushima Medical University, Department
Locations (1):
- Fukushima Medical University Hospital, Fukushima, Fukushima, Japan

REFERENCES:
- [Background] Niethammer AG, Xiang R, Becker JC, Wodrich H, Pertl U, Karsten G, Eliceiri BP, Reisfeld RA. A DNA vaccine against VEGF receptor 2 prevents effective angiogenesis and inhibits tumor growth. Nat Med. 2002 Dec;8(12):1369-75. doi: 10.1038/nm1202-794. Epub 2002 Nov 4. PMID 12415261
- [Background] Ishizaki H, Tsunoda T, Wada S, Yamauchi M, Shibuya M, Tahara H. Inhibition of tumor growth with antiangiogenic cancer vaccine using epitope peptides derived from human vascular endothelial growth factor receptor 1. Clin Cancer Res. 2006 Oct 1;12(19):5841-9. doi: 10.1158/1078-0432.CCR-06-0750. PMID 17020992
- [Background] Wada S, Tsunoda T, Baba T, Primus FJ, Kuwano H, Shibuya M, Tahara H. Rationale for antiangiogenic cancer therapy with vaccination using epitope peptides derived from human vascular endothelial growth factor receptor 2. Cancer Res. 2005 Jun 1;65(11):4939-46. doi: 10.1158/0008-5472.CAN-04-3759. PMID 15930316